CLINICAL TRIAL: NCT00118937
Title: Effect of Metformin On Glycaemic Control and Non-Glycaemic Cardiovascular Risk-Factors in Patients With Type-1 Diabetes, With Long-Standing Inadequate Glycaemic Control by Insulin and Diet
Brief Title: Effect of Metformin in Patients With Type-1 Diabetes With Inadequate Glycaemic Control by Insulin and Diet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Type-1-Metformin
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Placebo Comparator): Single-blind placebo run-in period. Duration one month.
  Interventions: Drug: Placebo.
- 2 (Active Comparator): Metformin 2000 mg, double-masked randomized during 12 months.
  Interventions: Drug: Metformin
- 3 (Placebo Comparator): Placebo, double-masked randomized during 12 months.
  Interventions: Drug: Placebo.

INTERVENTIONS:
Drug: Metformin — Tablet Metformin 500 mg, Dosage: 1000 mg two times daily (2000 mg total daily dose).
  Arms: 2
Drug: Placebo. — Tablet Placebo (corresponding to 500 mg metformin). Dosage: 1 tablet per day.
  Arms: 1
Drug: Placebo. — Tablet Placebo (corresponding to 500 mg metformin). Dosage: 2 tablets two times daily.
  Arms: 3

SUMMARY:
Ninety percent of patients with type-1-diabetes will develop late-diabetic complications in the eyes, kidneys, nervous- or cardiovascular-system. Poor glycaemic control is an important risk-factor for development of these late-diabetic complications. The Diabetes Control and Complications Trial (DCCT)-study showed, that improved glycaemic control can prevent the development and progression of these late-diabetic complications. Until now treatment with insulin- and diet-therapy has been the only treatment-modalities available to improve the glycaemic control in patients with type-1-diabetes. A substantial number of these patients still have long-standing poor glycaemic control despite intensive treatment with insulin- and diet-therapy.

The antidiabetic drug metformin has shown to be able to improve the glycaemic control in combination with insulin and furthermore reduce both mortality and the risk of developing cardiovascular disease in patients with type-2-diabetes.

Only few small studies have investigated the effect of treatment with metformin in patients with type-1-diabetes. These studies have suggested a positive effect of metformin in these patients too.

Method:

100 patients with type-1-diabetes with persistent poor glycaemic control i.e. HbA1c > 8.5% during the last 12 months are eligible. Patients are treated for one month with placebo. Hereafter half of the patients will be treated with metformin and the other half continues with placebo for 12 months both as add-on therapy. All patients are continuing ongoing treatment with insulin throughout the study. Before and after the start of treatment with metformin the effect on glycaemic control and other known risk-factors for development of cardiovascular disease i. e. blood-pressure, fasting lipids, urine-albumine-excretion, endothelial dysfunction, inflammation, fibrinolysis etc. is assessed.

This study will show if treatment with metformin can improve the glycaemic control and hereby the prognosis of patients with type-1-diabetes with persistent poor glycaemic control despite intensive treatment with insulin- and diet-therapy. This group of patients suffers the highest risk of developing late-diabetic complications with reduced quality of life and life-expectancy as a consequence.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c > 8.5% for more than one year prior to enrolment.
* Diabetes-duration > 5 years.
* Age at onset of diabetes < 35 years
* Fasting C-peptide < 300 pmol/l
* Age > 18 years at enrolment.

Exclusion Criteria:

* Clinical or biochemical signs of kidney-, liver- or heart-failure.
* Other coexisting serious morbidity, which will affect the study-participation or outcome of the study i.e. cancer.
* Known abuse of any medication or alcohol
* Hypoglycaemia unawareness.
* Pregnancy or planned pregnancy in the study-period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-12; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
HbA1c - difference between final visit and baseline.

SECONDARY OUTCOMES:
Absolute HbA1c
Number of mild and severe hypoglycaemia with or without measurements of blood-glucose.
Insulin-dose
The following parameters are measured at baseline and at the final visit after 12 months of intervention:
Plasma-PAI-antigen and -activity, t-PA-antigen- and activity.
Plasma-fibrinogen
Serum-albumin
Markers of endothelial dysfunction: Von Willebrand Factor, ICAM, VCAM, Amadori-protein, selectin and endothelin.
Plasma-homocysteine
Asymmetric DiMethylArginine - ADMA
Urine-albumin-excretion in three 24 hour urine-collections
Blood-pressure in the sitting position after 10 minutes of rest.
Fasting lipid-profile (total-cholesterol, LDL-cholesterol, HDL-cholesterol, VLDL-cholesterol and triglycerides), small-dense-LDL, Lp(a) and Apo-B100.
Weight, BMI and Waist-hip-ratio
White blood-cell-count, hs-CRP, Interleukin-6 and TNF-alfa.
Serum-creatinine, sodium, potassium, ASAT, alkaline phosphatase, Factor 2, 7, 10, Cobalamin, Erythrocyte-folate and Haemoglobin-concentration.
Extra blood- and urine-samples will be stored at -80 degrees Celsius for potential extra analyses after closure of the study. DNA will be stored for later pharmaco-genetic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Allan A Vaag, M.D., chief physician, Study Chair — Steno Diabetes Center Copenhagen; Soeren S Lund, M. D., Principal Investigator — Steno Diabetes Center Copenhagen

REFERENCES:
- [Derived] Lund SS, Tarnow L, Astrup AS, Hovind P, Jacobsen PK, Alibegovic AC, Parving I, Pietraszek L, Frandsen M, Rossing P, Parving HH, Vaag AA. Effect of adjunct metformin treatment in patients with type-1 diabetes and persistent inadequate glycaemic control. A randomized study. PLoS One. 2008;3(10):e3363. doi: 10.1371/journal.pone.0003363. Epub 2008 Oct 9. PMID 18852875